CLINICAL TRIAL: NCT00095108
Title: A Phase 1 Open-Label Study of the Safety and Pharmacokinetics of Recombinant Human Interleukin-21 (rIL-21) in Subjects With Metastatic Melanoma or Metastatic Renal Cell Carcinoma
Brief Title: Study of Interleukin-21 for Metastatic Malignant Melanoma and Metastatic Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ZymoGenetics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 494C10
Record Dates: First submitted 2004-10-29; First posted 2004-11-01 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Melanoma; Kidney Neoplasms; Metastases
Keywords: Metastatic Melanoma; Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Melanoma; Kidney Neoplasms; Neoplasm Metastasis; Carcinoma, Renal Cell

INTERVENTIONS:
Drug: Recombinant Human Interleukin-21

SUMMARY:
This study is being done to see if an experimental drug called recombinant interleukin-21 (rIL-21) when given to patients with stage 4 malignant melanoma or stage 4 kidney cancer is safe and has any effect on these types of cancers.

DETAILED DESCRIPTION:
This is a phase 1 safety study. Everyone enrolled and eligible will be given rIL-21. The study has 2 parts, Part A will determine how high a dose of rIl-21 can be safely given to patients with these types of cancers. Part B will determine if the drug is of any benefit to patients with these types of cancers. Part A may have up to 7 different dose groups. Beginning with the lowest dose, 3 patients will be treated and will be watched for side effects. If the side effects are not severe, the next group of 3 patients will recieve a higher dose. This cycle is repeated until the highest tolerated dose group is found.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older with stage 4 metastatic malignant melanoma or stage 4 metastatic kidney cancer
* ECOG status of 0 or 1
* Patients must have adequate liver, kidney and bone marrow function

Exclusion Criteria:

* Known ocular melanoma
* Suspected or confirmed brain metastases
* Patient cannot have had a bone marrow transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-05; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of rIL-21
To further characterize the safety of rIL-21 at the MTD

SECONDARY OUTCOMES:
Characterize pharmacokinetics of rIL-21
Evaluate immunogenicity of rIL-21
Identify clinical or biological parameters that may correlate with clinical efficacy
Characterize anti-tumor effect of IL-21

CONTACTS AND LOCATIONS:
Overall Officials: Diana Hausman, MD, Study Director — ZymoGenetics
Locations (2):
- United States (2):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington